CLINICAL TRIAL: NCT01718821
Title: Assessments on Current Pain Managements in Upper Gastrointestinal Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Hsu-chih Chien, Doctoral student, National Cheng Kung University
Other Study IDs: A-ER-101-134
Record Dates: First submitted 2012-10-16; First posted 2012-10-31 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Pain; Neuropathic Pain; Depression; Quality of Life; Upper GI Cancer
MeSH Terms: conditions — Pain; Neuralgia; Depression; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced upper GI cancer patients: Upper GI cancers include: esophageal cancer, gastric cancer, ampulla vater cancer, pancreatic cancer and cholangiocarcinoma.

SUMMARY:
Pain is one of the most common symptoms associated with cancer. The approach to pain management compresses routine pain assessments, utilizes both pharmacologic and nonpharmacologic interventions, and requires ongoing reevaluation of the patient. Cancer pain can be well controlled in the vast majority of patients if the algorithms of pain control are systematically applied, carefully monitored, and tailored to the needs of the individual patient.This study is aimed to assess the current pain managements in upper gastrointestinal cancer patients in Taiwan. The effects of neuropathic pain and depression on the enrolled patients would also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnose of advanced upper GI cancer based on pathology or imaging studies
* could report pain intensities and answer questionnaires by him/herself

Exclusion Criteria:

* with major neurologic or psychiatric diseases
* could not report pain intensities and answer questionnaires by him/herself

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients or out patients in National Cheng Kung University Hospital (a medical center)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain, assessed by BPI-SF. | Assessed at enrolled date (Day 1)
  Pain intensities of participants would be assessed by BPI-SF at D1.
Changes in pain, assessed by BPI-SF. | Baseline and 1 month.
  Changes in pain intensities of participants would be assessed by BPI-SF. The changes in pain would be assessed again after 1 month when participants have outpatient visits or during their admission. An expected following duration average of would be 4 weeks.

SECONDARY OUTCOMES:
Depression, assessed by two stem questions. | Assessed at enrolled date (Day 1)
  Depression of participants would be assessed by questionnaires as mentioned at D1.
Changes in depression, assessed by two stem questions. | Baseline and 1 month.
  Changes in depression status would be assessed by questionnaires as mentioned. The changes would be assessed again after 1 month when participants have outpatient visits or during their admission. An expected following duration average of would be 4 weeks.
Quality of life, assessed by EROTC QLQ C30. | Day 1
  Quality of life of participants would be assessed by questionnaires as mentioned at D1.
Neuropathic pain, assessed by DN4 questions. | Day 1
  Neuropathic pain of participants would be assessed by questionnaires as mentioned at D1.
Changes in quality of life. Quality of life, assessed by EROTC QLQ C30. | Baseline and 1 month.
  Changes in quality of life would be assessed by questionnaires as mentioned. The changes would be assessed again after 1 month when participants have outpatient visits or during their admission. An expected following duration average of would be 4 weeks.
Changes in neuropathic pain. Neuropathic pain, assessed by DN4 questions. | Baseline and 1 month.
  Changes in neuropathic pain would be assessed by questionnaires as mentioned. The changes would be assessed again after 1 month when participants have outpatient visits or during their admission. An expected following duration average of would be 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yea-huei Kao Yang, Principal Investigator — Institute of Clinical Pharmacy and Pharmaceutical Science, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Tainan, Taiwan